CLINICAL TRIAL: NCT05247320
Title: Prospective Evaluation Analysis and Kinetics of IV Sotalol
Brief Title: Prospective Evaluation Analysis and Kinetics Registry
Acronym: PEAKS
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: AltaThera Pharmaceuticals, LLC (Unknown)
Responsible Party: Principal Investigator, Benjamin A. Steinberg, Associate Professor, University of Utah
Other Study IDs: 00147440
Record Dates: First submitted 2022-01-07; First posted 2022-02-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Atrial Arrhythmia
Keywords: Atrial Arrhythmia; Sotalol
MeSH Terms: interventions — Sotalol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective
  Interventions: Drug: Sotalol Injection
- Retrospective
  Interventions: Drug: Sotalol Injection

INTERVENTIONS:
Drug: Sotalol Injection — Standard of care IV sotalol infusion for atrial arrhythmias

SUMMARY:
In a cohort of patients electively treated for atrial arrhythmia with IV sotalol (initiation or dose escalation), this study will describe patient characteristics, short-term safety and efficacy, electrocardiographic monitoring, and PK and PD parameters (in a subset) associated with IV dosing approach.

DETAILED DESCRIPTION:
Antiarrhythmic drug therapy plays a vital role in the achievement of rhythm control in patients with atrial arrhythmias. Class III antiarrhythmic drugs are frequently used in these patients. However, these drugs are associated with a nontrivial risk of QT interval prolongation and associated risk of life-threatening ventricular arrhythmias. In this setting, initiation and dose titration of these drugs is often performed on an inpatient basis for the first five oral doses, typically requiring hospitalization for two days or longer.

The availability of sotalol in intravenous (IV) form, recently approved for initiation or dose increase among patients with atrial arrhythmias, affords an opportunity to shorten hospitalization for these patients. This approach was approved based on translational science research that used computer-based simulation modeling to predict sotalol concentrations. There remain knowledge gaps regarding the use of IV sotalol in these patients, specifically around real-world outcomes, as well as pharmacodynamic and pharmacokinetic profiles in patients. The purpose of this registry is to collect data among patients and centers using IV sotalol loading for initiation or dose titration in the treatment of atrial arrhythmias, in order to fill the above knowledge gaps.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years and older
2. Eligible for the use of elective intravenous sotalol loading to treat atrial arrhythmias, per the treating clinician
3. IV sotalol infusion started for the treatment of atrial arrhythmias, in the setting of initiation or dose titration of chronic sotalol therapy
4. Elective hospital admission primarily for loading with intravenous sotalol with/without cardioversion, with no other planned therapy or procedures

Exclusion Criteria:

1. Study materials not available in the subject's preferred language.
2. Patients undergoing treatment for active concomitant ventricular arrhythmias
3. Standard exclusions for elective sotalol use (at the time of initiation):

   * Heart rate < 40 bpm or 2nd/3rd degree AV block without pacemaker
   * QTc ≥ 450 in absence of bundle branch block (≥ 500 in the presence of a bundle branch block)
   * Severe left ventricular hypertrophy (thickness >1.5 cm)
4. Patients who were previously intolerant to antiarrhythmic class III therapy
5. Patients missing key data elements in their electronic health record (for retrospective subjects only).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry study will enroll adult patients 18 years and older electively treated for atrial arrhythmia with standard of care IV sotalol (initiation or dose escalation). During their elective hospitalization the patient is not planned to receive any other intervention. The registry allows retrospective and prospective enrollment. Patients will be excluded if they are undergoing treatment for active concomitant ventricular arrhythmias, intolerant to class III antiarrhythmic therapy, not meeting standard criteria to receive elective IV sotalol, or if key data elements not available (retrospective enrolled patients only). Approximately 150 patients will be enrolled and for about 20 patients PK/PD data will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants completing IV sotalol loading for atrial arrhythmias | Enrollment of patient until 7 days following discharge
  To describe the characteristics of patients receiving treatment for atrial arrhythmias with the IV formulation of Sotalol.

SECONDARY OUTCOMES:
Number of participants with symptomatic/actionable bradycardia. | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with QTc prolongation >500 ms (or 550 ms for underlying BBB). | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with recurrent AT/AF +/- RVR. | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with any ventricular arrhythmia (sustained or non-sustained. | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with Sudden Cardiac Death (SCD) (including aborted). | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with Hypotension Symptomatic or <=90/50. | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with unplanned hospitalization prolongation. | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with unplanned rehospitalization. | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.
Number of participants with death. | Infusion IV Sotalol out to 3 months.
  To describe the short-term safety and efficacy outcomes among patients receiving IV Sotalol for atrial arrhythmias in clinical practice.

OTHER OUTCOMES:
Sotalol levels measured at 0-30 minutes before IV dose. | 0 - 30 min before IV dose
  To describe the pharmacokinetics (PK) of IV Sotalol in vivo and compare it to the profiles predicted through modeling.
Sotalol levels measured at 0-5 minutes after end of IV infusion. | 0-5 minutes after end of IV infusion.
  To describe the pharmacokinetics (PK) of IV Sotalol in vivo and compare it to the profiles predicted through modeling.
Sotalol levels measured at 3 hours ± 5 minutes after end of IV infusion. | 3 hours ± 5 minutes after end of IV infusion.
  To describe the pharmacokinetics (PK) of IV Sotalol in vivo and compare it to the profiles predicted through modeling.
Sotalol levels measured at 0-30 minutes before first enteral dose. | 0-30 minutes before first enteral dose.
  To describe the pharmacokinetics (PK) of IV Sotalol in vivo and compare it to the profiles predicted through modeling.
Sotalol levels measured at 2-4 hours after second enteral dose. | 2-4 hours after second enteral dose.
  To describe the pharmacokinetics (PK) of IV Sotalol in vivo and compare it to the profiles predicted through modeling.
Sotalol levels measured at 2-4 hours after first enteral dose. | 2-4 hours after first enteral dose.
  To describe the pharmacokinetics (PK) of IV Sotalol in vivo and compare it to the profiles predicted through modeling.
Number of participants on outpatient, mobile ECG with Bradycardia <= 40 bpm. | Enrollment until 7 days following discharge
  Assess the use of mobile ECG to detect clinically-significant arrhythmia and changes to heart rate and QTc among these patients.
Number of participants on outpatient, mobile ECG with recurrent AT/AF +/- RVR. | Enrollment until 7 days following discharge
  Assess the use of mobile ECG to detect clinically-significant arrhythmia and changes to heart rate and QTc among these patients.
Number of participants on outpatient, mobile ECG with QTc prolongation >500 ms (or 550 ms for underlying BBB). | Enrollment until 7 days following discharge
  Assess the use of mobile ECG to detect clinically-significant arrhythmia and changes to heart rate and QTc among these patients.
Number of participants on outpatient, mobile ECG with any ventricular arrhythmia (sustained or non-sustained). | Enrollment until 7 days following discharge
  Assess the use of mobile ECG to detect clinically-significant arrhythmia and changes to heart rate and QTc among these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A. Steinberg, MD, MHS, Principal Investigator — University of Utah; Jonathan Pinccini, MD, Principal Investigator — Duke University; Suneet Mittal, MD, Principal Investigator — Valley Health; Parash Pokharel, MD, Principal Investigator — Geisinger Health; Thomas F Deering, MD, Principal Investigator — Piedmont Heart Institute; Robert Kennedy, MD, Principal Investigator — Munson Medical Center; Michael West, MD, Principal Investigator — Presbyterian Healthcare Services; Sergio Cossu, MD, Principal Investigator — Lehigh Valley Health Network; Nishant Verma, MD, Principal Investigator — Northwestern University; Jonathan Silver, MD, Principal Investigator — Lahey Hospital & Medical Center; Abhishek Deshmukh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Somberg JC, Vinks AA, Dong M, Molnar J. Model-Informed Development of Sotalol Loading and Dose Escalation Employing an Intravenous Infusion. Cardiol Res. 2020 Oct;11(5):294-304. doi: 10.14740/cr1143. Epub 2020 Aug 7. PMID 32849964
- [Background] Samanta R, Thiagalingam A, Turner C, Lakkireddy DJ, Kovoor P. The Use of Intravenous Sotalol in Cardiac Arrhythmias. Heart Lung Circ. 2018 Nov;27(11):1318-1326. doi: 10.1016/j.hlc.2018.03.017. Epub 2018 Mar 29. PMID 29853342
- [Background] Somberg JC, Preston RA, Ranade V, Molnar J. QT prolongation and serum sotalol concentration are highly correlated following intravenous and oral sotalol. Cardiology. 2010;116(3):219-25. doi: 10.1159/000316050. Epub 2010 Aug 7. PMID 20693799
- [Background] Von Bergen NH, Beshish AG, Maginot KR. Outpatient intravenous sotalol load to replace 3-day admission oral sotalol load. HeartRhythm Case Rep. 2019 Apr 24;5(7):382-383. doi: 10.1016/j.hrcr.2019.04.005. eCollection 2019 Jul. No abstract available. PMID 31341782
- [Background] Etheridge SP, Asaki SY. An Exciting New Tool in the Electrophysiologist's Toolbox, Intravenous Sotalol: Faster, Safer, Better? JACC Clin Electrophysiol. 2020 Apr;6(4):433-435. doi: 10.1016/j.jacep.2019.12.016. No abstract available. PMID 32327077
- [Derived] Steinberg BA, Mittal S, Holubkov R, Groh CA, Kennedy R, Pokharel P, Perez M, Savona SJ, Verma N, Watt K, Piccini JP, Bunch TJ, Deering TF. Correlation between mobile and 12-lead ECG among patients loading with intravenous sotalol: A PEAKS substudy. Heart Rhythm O2. 2025 Feb 11;6(4):499-508. doi: 10.1016/j.hroo.2025.01.018. eCollection 2025 Apr. PMID 40321743
- [Derived] Steinberg BA, Holubkov R, Bunch TJ, Deering TF, Groh CA, Kennedy R, Perez M, Piccini JP, Pokharel P, Savona SJ, Verma N, Watt K, Mittal S. Sotalol Dosing and Outcomes Among Patients Undergoing Intravenous Loading for Atrial Arrhythmias-A PEAKS Registry Substudy. J Cardiovasc Electrophysiol. 2025 Jun;36(6):1352-1358. doi: 10.1111/jce.16677. Epub 2025 Apr 9. PMID 40205819